CLINICAL TRIAL: NCT03095560
Title: Role of Body Shadow in Improving Virtual Reality Rehabilitation: Preliminary Data From BTS Nirvana
Brief Title: BTs Nirvana and Post-stroke Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Principal investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSVR
Record Dates: First submitted 2017-03-18; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Virtual Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-immersive virtual training with shadow (S-IVTS) (Experimental): All the participants underwent a neurocognitive-rehabilitative training consisting of 24 sessions of BTsN. Each treatment session lasted 45 minutes, and was repeated three times a week for 8 weeks. in the BTsN device used in the S-IVTS group the projector is located behind the patient, thus the shadow of the patient is projected on the screen.
  Interventions: Device: NIRVANA
- Semi-immersive virtual training without shadow (S-IVT) (Experimental): All the participants underwent a neurocognitive-rehabilitative training consisting of 24 sessions of BTsN. Each treatment session lasted 45 minutes, and was repeated three times a week for 8 weeks. in the BTsN device used in the S-IVT group the projector is located in front of the patient and the shadow is not visible.
  Interventions: Device: NIRVANA

INTERVENTIONS:
Device: NIRVANA — Nirvana is the first device based on optoelectronic infrared sensors, though which the patient can simply interact through his movements. The rehabilitation exercises with audio-visual stimuli and feedback involve the perceptual-cognitive skills of patients, resulting in a motivational training. Several modes and increasing levels of difficulty characterize each exercise, so the therapist can use a pre-defined rehabilitative solution or new ones, according to patient's needs. The results achieved during rehabilitation allow the therapist to evaluate the patient's actual progress, and then to modify the rehabilitation program. The system is connected to a projector or a big screen (put in front of the patient), reproducing an interactive series of exercises (for trunk, upper and lower limbs, and cognition), thanks to an infrared video camera analyzing the patient's movements, it creates interactivity.

SUMMARY:
Purpose of the article: aim of the present study was to detect the differences between the presence or not of body shadows during a virtual reality (VR) training with BTS NIRVANA (BTsN). Materials and methods: In this pilot study, we enrolled 20 post-stroke rehabilitation inpatients, who underwent a neurocognitive-rehabilitative training consisting of 24 sessions (three times a week for 8 weeks) of BTsN. All the patients were randomized into two groups: Semi-immersive virtual training with (S-IVTSgroup) or without (S-IVTgroup) body shadows.

Each participant was evaluated before (T0), and immediately (T1) after the end of the training by a skilled neuropsychologist through the administration of a complete battery, and by a skilled neurologist to assess motor functions.

DETAILED DESCRIPTION:
In this pilot study, we enrolled 20 post-stroke rehabilitation inpatients, who attended the Laboratory of Robotic and Cognitive Rehabilitation of IRCCS Neurolesi of Messina from June 2016 to January 2017. The inclusion criteria were: ischemic or hemorrhagic stroke in the chronic phase (i.e., at least 6 months from the acute neurological event); inability to stand independently for more than one minute; ability to sit for at least 20 minutes (including at least one minute without support); presence of moderate to mild cognitive impairment (Mini-Mental State Examination from 10 to 23); absence of disabling sensory alterations, severe psychiatric and other medical illness. The study was approved by the Local Ethical Committee. All the patients, adequately informed about the study, offered their collaboration, and provided informed consent to enter the study. All the participants underwent a neurocognitive-rehabilitative training consisting of 24 sessions of BTsN. Each treatment session lasted 45 minutes, and was repeated three times a week for 8 weeks. Both the groups underwent the same conventional physiotherapy program. All the patients were randomized into two groups: Semi-immersive virtual training with (S-IVTSgroup) or without (S-IVTgroup) body shadows.

Each participant was evaluated by a skilled neuropsychologist through the administration of a complete battery, and by a skilled neurologist to assess motor functions. All the patients were evaluated by a specific clinical-psychometric battery before (T0), and immediately (T1) after the end of the training. Primary outcomes consisted of the Montreal Cognitive Assessment Test (MoCA) and the Functional Independence Measure (FIM). In addition, we administered the Frontal Assessment Battery (FAB) to assess executive functions, Attentive Matrices (AM) and Trial Making Test (TMTA, TMTB, and TMTB-A) to measure the attention process, and the Trunk Control Test (TCT) and Motricity Index (MI) for upper limbs to evaluate motor functions.

BTsN TRAINING SETTING Nirvana is the first device based on optoelectronic infrared sensors, though which the patient can simply interact through his movements. The rehabilitation exercises with audio-visual stimuli and feedback involve the perceptual-cognitive skills of patients, resulting in a motivational training. Several modes and increasing levels of difficulty characterize each exercise, so the therapist can use a pre-defined rehabilitative solution or new ones, according to patient's needs. The results achieved during rehabilitation allow the therapist to evaluate the patient's actual progress, and then to modify the rehabilitation program. The system is connected to a projector or a big screen (put in front of the patient), reproducing an interactive series of exercises (for trunk, upper and lower limbs, and cognition), thanks to an infrared video camera analyzing the patient's movements, it creates interactivity. At the end of each work session, it is possible to export the full list of all exercises performed and the score obtained for each of them. Concerning cognitive training, we included a series of exercises involving attention, memory (verbal and visuo-spatial), spatial cognition, ocular-manual coordination, gnosis abilities, problem solving, executive function, and constructive praxis.

Notably, in the BTsN device used in theS-IVT group the projector is located behind the patient, thus the shadow of the patient is projected on the screen, whereas in the S-IVTSgroup the projector is located in front of the patient and the shadow is not visible.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were: ischemic or hemorrhagic stroke in the chronic phase (i.e., at least 6 months from the acute neurological event); inability to stand independently for more than one minute; ability to sit for at least 20 minutes (including at least one minute without support); presence of moderate to mild cognitive impairment (Mini-Mental State Examination from 10 to 23);

Exclusion Criteria:

* absence of disabling sensory alterations, severe psychiatric and other medical illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment Test (MoCA) | Six months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Russo M, De Luca R, Naro A, Sciarrone F, Aragona B, Silvestri G, Manuli A, Bramanti A, Casella C, Bramanti P, Calabro RS. Does body shadow improve the efficacy of virtual reality-based training with BTS NIRVANA?: A pilot study. Medicine (Baltimore). 2017 Sep;96(38):e8096. doi: 10.1097/MD.0000000000008096. PMID 28930852